CLINICAL TRIAL: NCT07171281
Title: Precise Eating Time to Improve Glycemic Control and Cardiometabolic Health in Prediabetes and Diabetes: the GLYCOTIME Trial
Brief Title: Precise Eating Time to Improve Glycemic Control and Cardiometabolic Health in Prediabetes and Diabetes
Acronym: GLYCOTIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: Technische Universität Dresden, Germany (Unknown); University of Surrey, UK (Unknown); University of Geneva, Switzerland (Other); Technische Universität München, Germany (Unknown); German Diabetes Center (DDZ), Germany (Unknown); University of Rovira i Virgili, Spain (Unknown)
Responsible Party: Principal Investigator, Olga Ramich (formerly Pivovarova), Head of Department Molecular Metabolism and Precision Nutrition, German Institute of Human Nutrition
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 85/2023; TEMP643937-BO-ff (Other: Ethics committee LAEKB)
Record Dates: First submitted 2025-08-26; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Prediabetes; Type 2 Diabetes; Obesity &Amp; Overweight
Keywords: Time-restricted eating; Prediabetes; Type 2 Diabetes; Chrononutrition; Glucose metabolism; Overweight; Obesity; Continuous glucose monitoring; TRE; Prevention and treatment of type 2 diabetes
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2; Obesity; Overweight; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Time-Restricted Eating (Experimental)
  Interventions: Behavioral: Early Time-Restricted Eating
- Late Time-Restricted Eating (Experimental)
  Interventions: Behavioral: Late Time-Restricted Eating

INTERVENTIONS:
Behavioral: Early Time-Restricted Eating — Participants will restrict their eating window (8 hours eating and 16 hours fasting per day) and caloric intake moderately.
  During the early TRE intervention, participants will primarily consume their meals in the morning. The precise eating window will be defined based on the individual chronotype of the participants. Additionally, participants will be required to reduce their daily caloric consumption by 25%. They will replace one daily meal with a calorie-reduced product to facilitate caloric restriction.
  Other Names: eTRE; early TRE
  Arms: Early Time-Restricted Eating
Behavioral: Late Time-Restricted Eating — Participants will restrict their eating window (8 hours eating and 16 hours fasting per day) and caloric intake moderately.
  During the late TRE intervention, participants will primarily consume their meals in the evening. The precise eating window will be defined based on the individual chronotype of the participants. Additionally, participants will be required to reduce their daily caloric consumption by 25%. They will replace one daily meal with a calorie-reduced product to facilitate caloric restriction.
  Other Names: LateTRE; lTRE
  Arms: Late Time-Restricted Eating

SUMMARY:
The objective of this study is to investigate the impact of hypocaloric time-restricted eating (TRE) at different day times (early versus late TRE) on glucose metabolism and other cardiometabolic parameters in individuals with overweight and with normal, or impaired glucose metabolism (prediabetes and type 2 diabetes). In addition, the study aims to elucidate the molecular mechanisms underlying these effects.

DETAILED DESCRIPTION:
This dietary intervention study will follow a crossover design. During the intervention phases, participants will restrict their dietary intake to a defined eating window of 8 hours - predominantly in the morning (early TRE) or predominantly in the afternoon (late TRE) - in conjunction with a moderate caloric restriction for five weeks. A 10-12-week washout phase will separate the intervention periods.

Overweight and obese individuals with healthy glucose metabolism, prediabetes, or non-insulin-treated type 2 diabetes will be recruited for the study.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obesity (BMI 25-40 kg/m²)
* Healthy glucose metabolism (fasting glucose <100 mg/dl and glucose after 2 hours OGTT <140 mg/dl)
* OR impaired glucose metabolism (fasting glucose 100-125 mg/dl and/or glucose after 2 hours OGTT 140-199 mg/dl and/or HbA1c 5.7-6.4%)
* OR type 2 diabetes (according to existing medical diagnosis or fasting glucose >126 mg/dl and/or glucose after 2 hours OGTT >200 mg/dl and/or HbA1c ≥6.5%)
* Daily eating window ≥12 hours

Exclusion Criteria:

* Weight changes > 5% within past 3 months
* Shift work
* Traveling across more than one time zone within one month prior to the study
* Pregnancy and breastfeeding
* Eating disorders, food intolerance/allergy to ingredients in the diet product, vegan diet, practicing time-restricted eating
* Severe chronic illnesses or other conditions that are incompatible with the planned intervention and examination program (e.g. type 1 diabetes, recent cardiovascular event, malabsorption, cancer in the last two years, etc.)
* Treatment with insulin, sulfonylureas, and GLP-1 receptor agonists, steroid use (oral, cutaneous, or parenteral), regular intake of melatonin, anticoagulation treatment that cannot be paused
* Extreme early and extreme late chronotypes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-19 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Mean 24-hour glucose | 5 weeks
  Mean 24-hour glucose assessed by continuous glucose monitoring (CGM)

SECONDARY OUTCOMES:
Glycemic variability | 5 weeks
  Inter- and intraday indices of glycemic variability assessed by CGM
Glucose levels | 5 weeks
  Fasting and postprandial glucose [mg/dL] in response to a mixed meal tolerance test
Insulin levels | 5 weeks
  Fasting and postprandial insulin [mU/L] in response to a mixed meal tolerance test
Glucagon levels | 5 weeks
  Fasting and postprandial glucagon [pmol/L] in response to a mixed meal tolerance test
Insulin resistance | 5 weeks
  Insulin resistance, as assessed by HOMA-IR [AU]
Insulin secretion | 5 weeks
  Insulin secretion, as assessed with the insulinogenic index [AU]
Body weight | 5 weeks
  Body weight [kg], as measured by scale weight
Body Mass Index (BMI) | 5 weeks
  BMI [kg/m2], calculated as weight/square height
Waist and hip circumference | 5 weeks
  Waist and hip circumference [cm] measured by tape
Body composition | 5 weeks
  Body fat mass and lean mass [kg], as measured by bioelectrical impendance analysis (BIA)
Fasting cholesterol | 5 weeks
  Fasting total cholesterol, low-density lipoprotein and high-density lipoprotein cholesterol [mmol/L]
Fasting triglycerides | 5 weeks
  Fasting triglycerides [mmol/L]
Blood pressure | 5 weeks
  Systolic and diastolic blood pressure [mm Hg], as measured by manometer
Resting energy expenditure | 5 weeks
  Resting energy expenditure [kcal/day], as assessed by indirect calorimetry
Gene expresssion in adipose tissue | 5 weeks
  RNAseq analysis of subcutaneous adipose tissue samples
Inflammatory markers in blood and adipose tissue | 5 weeks
  Levels of adipokines and inflammatory markers measured in blood samples and subcutaneous adipose tissue samples
Subjective satiety and hunger sensation | 5 weeks
  Satiety and hunger scores assessed using Visual Analog Scales (VAS, with a scale of 1-100, where higher values correspond to stronger satiety/hunger)
Concentration of satiety and hunger regulating hormones | 5 weeks
  Levels of ghrelin and peptide YY (PYY), as measured in blood samples in [pg/mL]
Species and strain-level microbiome changes | 5 weeks
  Species and strain-level microbiome changes, as assessed by 16S rRNA gene sequencing of stool samples
Levels of microbiome-derived metabolites | 5 weeks
  Levels of microbiome-derived metabolites measured in stool samples and blood plasma
Sleep quality | 5 weeks
  Sleep quality as assessed by the Pittsburgh Sleep Quality Index (PSQI score, which ranges from 0-21, where higher values correspond to worse sleep quality) and also monitored by an ActiGraph device
Sleep and wake timing | 5 weeks
  Sleep onset and offset assessed by the Pittsburgh Sleep Quality Index (PSQI score, which ranges from 0-21, where higher values correspond to worse sleep quality) and in addition by using a sleep diary
Internal circadian phase | Screening visit (week 0)
  Internal circadian phase as assessed using the BodyTime assay in peripheral mononuclear blood cells (PBMCs)
Glucagon-like peptide-1 levels | 5 weeks
  Fasting and postprandial glucagon-like peptide-1 (GLP-1) in response to a mixed meal tolerance test [pM]
Gastric inhibitory polypeptide | 5 weeks
  Fasting and postprandial gastric inhibitory polypeptide (GIP) in response to a mixed meal tolerance test [pg/mL]
Gene expresssion in peripheral mononuclear blood cells (PBMCs) | 5 weeks
  RNAseq analysis of clock, metabolic and inflammatory gene expression peripheral mononuclear blood cells (PBMCs)
Malondialdehyde | 5 weeks
  Plasma malondialdehyde [µmol/L]
3-nitrotyrosine | 5 weeks
  Plasma 3-nitrotyrosine [pmol/mg]
Protein carbonyls | 5 weeks
  Plasma protein carbonyls [nmol/mg]
36-item Short Form Health Survey (SF-36) to measure health-related quality-of-life | 5 weeks
  Health-related quality-of-life, as assessed by the 36-Item Short Form Health Survey (SF-36, with scores ranging from 0 to 100, with a higher score defining a more favorable health state)
Satisfaction with the intervention | 5 weeks
  Satisfaction with the intervention assessed by a 5-point Likert scale (with 5 representing "Very satisfied" and 1 representing "Very dissatisfied")
Decision behavior | 5 weeks
  Impulsiveness assessed by decision making tasks on computer

OTHER OUTCOMES:
Physical activity level | 5 weeks
  24-h physical activity level (light, moderate, sedentary activity, metabolic equivalent of task) will be monitored by an Actigraph device
Liver enzyme levels and renal values | 5 weeks
  γ-glutamyltransferase (GGT), aspartate aminotransferase (ALT), and alanine aminotransferase (AST), creatinine, urea, uric acid determined in fasting blood samples
Food intake | 5 weeks
  Energy intake [kcal/day] assessed by food records
Macronutrient intake | 5 weeks
  Percentage of calories from fat, carbohydrates, protein, and fiber, determined based on dietary records
Food timing | 5 weeks
  Start and stop times of daily eating window and clock time of each daily meal intake assessed by food records

CONTACTS AND LOCATIONS:
Locations (1):
- German Institute of Human Nutrition Potsdam-Rehbruecke, Nuthetal, Germany

IPD SHARING:
Plan to Share IPD: No